CLINICAL TRIAL: NCT04775537
Title: OssiMend Bioactive Moldable in Posterolateral Instrumented Lumbar Fusion
Brief Title: OssiMend BA in Posterolateral Instrumented Lumbar Fusion
Status: Recruiting | Type: Observational
Sponsor: Collagen Matrix (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP.072.Spine Prospective
Record Dates: First submitted 2021-02-11; First posted 2021-03-01 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-01

CONDITIONS: Spinal Disease; Degenerative Disc Disease
Keywords: Bone Graft; Lumbar Fusion
MeSH Terms: conditions — Spinal Diseases; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- OssiMend™ Bioactive Moldable: Patients undergoing Lumber Spine Fusion
  Interventions: Device: OssiMend™ Bioactive Moldable

INTERVENTIONS:
Device: OssiMend™ Bioactive Moldable — Lumbar Spine fusion with OssiMend™ Bioactive Moldable

SUMMARY:
The primary objective of this study is to measure the success rate of lumbar fusion in subjects at 12 months when instrumented lumbar arthrodesis is performed using OssiMend Bioactive Moldable as the bone grafting material

DETAILED DESCRIPTION:
The primary objective of this study is to measure the success rate of lumbar fusion in subjects at 12 months when instrumented lumbar arthrodesis is performed using OssiMend Bioactive Moldable as the bone grafting material. The primary endpoints are radiographic evidence of fusion and the absence of serious adverse events attributable to OssiMend Bioactive Moldable. The secondary objective is to evaluate the clinical outcomes over a period of 1 year (2 years, if possible).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older at the time of consent and must have a documented diagnosis of degenerative disc disease (DDD) that has failed to respond to nonoperative treatment for at least 6 months. DDD is defined by back and/or radicular pain with degeneration of the disc as confirmed by medical history, physical examination, and radiographic studies that may include CT, MRI, plain X-ray film, discography, myelography, etc. with one or more of the following findings:

  * Instability as defined by >3mm translation or >5 degrees angulation
  * Osteophyte formation of facet joints or vertebral endplates
  * Decreased disc height, on average by >2mm, but dependent upon the spinal level
  * Herniated nucleus pulposus
  * Facet joint degeneration/changes

Exclusion Criteria:

1. Subject is under 18 years of age at the time of consent
2. Subject has had prior lumbar spine fusion surgery at any level
3. Subject is currently undergoing treatment for malignancy or has undergone treatment for malignancy
4. Subject is pregnant or nursing or planning to become pregnant during the two years (24 months) following arthrodesis
5. Subject has an active (local or systemic) infection or is undergoing adjunctive treatment for infection
6. Subjects under workers compensation or active litigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects must be 18 years of age or older at the time of consent and must have a documented diagnosis of degenerative disc disease (DDD) that has failed to respond to nonoperative treatment for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Fusion Success | 12 months
  Fusion will be assessed with A/P and Lateral radiographs taken and scored with Lenke's classification of posterolateral fusion success

SECONDARY OUTCOMES:
Visual analog scale (VAS) of back and leg (left and right) | 12 months
  Improvement of pain as defined by the Visual analog scale (VAS) of back and leg (left and right)
Oswestry Lower Back Pain Questionnaire | 12 months
  Pain/Disability as measured by Oswestry Lower Back Pain Questionnaire
SF36 | 12 months
  Pain and function as measured by the Short - Form 36

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - San Diego Neurosurgery, Encinitas, California
  - Hartford Hospital, Hartford, Connecticut
  - University Orthopaedic Associates, Division of OrthoNJ, Somerset, New Jersey
  - McKenzie-willamette Medical Center, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://collagenmatrix.com/